CLINICAL TRIAL: NCT06019442
Title: An Electronic Brief Intervention to Reduce Alcohol Consumption Intentions, Improve Alcohol Literacy, and Reduce Harmful Use Among Women Attending a Breast Screening Service: a Randomised Controlled Trial
Brief Title: An Electronic Brief Alcohol Intervention for Women Attending a Breast Screening Service (Health4Her)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turning Point (Other)
Collaborators: Monash University (Other); Eastern Health (Other); BreastScreen Victoria (Unknown); Lifepool (Unknown); Shades of Pink (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: LR22-071-91112
Record Dates: First submitted 2023-08-13; First posted 2023-08-31 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2023-12

CONDITIONS: Health Knowledge, Attitudes, Practice; Alcohol Drinking
Keywords: Women's health; Public health; Health promotion
MeSH Terms: conditions — Behavior; Alcohol Drinking | interventions — Ethanol; Methods

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial (2 arms) + pilot of modified active arm
  The pilot group does not form part of the planned randomised controlled trial or power and sample size calculation, but is included based on findings from the previous phase of this research (e.g. women not having time to complete the intervention onsite). Therefore n~20 women who cannot participate on the day of breast screening will be offered to participate in the modified active arm offsite.
Who Masked: Participant, Outcomes Assessor
Masking Description: The on-site researcher responsible for recruitment will not be blind to treatment assignment; the participating women self-completing baseline assessment, intervention, immediate post-intervention and 4-week follow-up assessments will be blinded to treatment assignment. The researcher who oversees follow-up assessment data collection will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief alcohol intervention (Health4Her-Automated) + lifestyle health promotion (Experimental): The intervention arm will receive:
  * brief alcohol intervention
  * lifestyle health promotion focused on physical activity and maintaining a healthy weight for reducing breast cancer risk.
  Participants will receive an iPad and earphones to self-complete the intervention. Alcohol and lifestyle information will be delivered by way of an animation on an iPad, and self-completed activities to reinforce intervention content.
  Interventions: Behavioral: Brief alcohol intervention (Health4Her-Automated); Behavioral: Lifestyle health promotion
- Lifestyle health promotion (Other): The control arm will receive:
  * lifestyle health promotion focused on physical activity and maintaining a healthy weight for reducing breast cancer risk.
  Participants will receive an iPad and earphones to self-complete the control intervention. Lifestyle information will be delivered by way of an animation on an iPad, and a self-completed activity to reinforce intervention content.
  Interventions: Behavioral: Lifestyle health promotion

INTERVENTIONS:
Behavioral: Brief alcohol intervention (Health4Her-Automated) — Embedded within the lifestyle health promotion provided in both conditions, participants randomised to the experimental condition will receive a brief alcohol intervention. The brief alcohol intervention will comprise information and behaviour-change content regarding alcohol consumption, including: messaging around alcohol risks/harms (with a focus on alcohol use and breast cancer risk), positive-framed messaging on the health benefits of reducing alcohol intake, and alcohol harm-reduction / behaviour change strategies (e.g. drink counting, goal setting, behaviour substitution, problem solving).
  Post-session information will be provided via email (i.e. electronic brochure summarising brief alcohol intervention content).
  Arms: Brief alcohol intervention (Health4Her-Automated) + lifestyle health promotion
Behavioral: Lifestyle health promotion — Lifestyle health promotion, focused on physical activity and maintaining a healthy weight for reducing breast cancer risk, will be provided.
  Post-session information will be provided via email (i.e. electronic brochure summarising nutrition for maintaining a healthy weight).

SUMMARY:
Alcohol is a major modifiable risk factor for female breast cancer; yet, awareness of this risk remains surprisingly low and is not systematically addressed in healthcare settings. This study aim to test the effectiveness of a co-designed, automated brief alcohol intervention (Health4Her-Automated) in reducing women's drinking intentions, improving alcohol literacy, and reducing consumption.

DETAILED DESCRIPTION:
Alcohol is a major modifiable risk factor for female breast cancer, even in very low amounts. In Australia, alcohol consumption accounts for 6.6 per cent of cases in post-menopausal women, and 18 per cent of breast cancer deaths. Yet, awareness of this risk remains low and is not systematically addressed in healthcare settings. Embedding a brief alcohol intervention within lifestyle information offered to all women attending breast screening provides the opportunity to address harmful drinking in a discrete, non-judgmental way, to prevent alcohol-attributable breast cancer among this at-risk population.

Brief alcohol interventions are short, single-session programs typically offered in general practice settings to gather information on a person's alcohol consumption and, in a non confrontational way, provide strategies and motivate change to reduce consumption and related risk of harm. An automated brief alcohol intervention, self-completed on a device such as an iPad, is a low-cost, labour- and time-efficient approach that overcomes many of the issues of providing intervention within busy healthcare environments.

Building on the previous pilot trial of a prototype brief e-health intervention (which included alcohol-related questions asked by a researcher, and an animation viewed on an iPad that was activated by the researcher), the aim of the current study is to test the effectiveness of a co-designed, automated brief alcohol intervention (Health4Her-Automated) in reducing women's drinking intentions, improving alcohol literacy, and reducing consumption.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 40+ years of age
* Attending routine breast screening
* With or without a breast cancer history
* Reporting any level of alcohol consumption

Exclusion Criteria:

* Not able to read or comprehend English to enable participation
* No access to a computer, tablet or smartphone to complete follow-up assessment
* Women who are pregnant (also an exclusion from breast screening)
* Participation in the pilot Health4Her trial

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Drinking intentions | immediately post-randomisation
  Change in next-month drinking intentions (5-point scale: 1, not at all; 5, to a very large extent)

SECONDARY OUTCOMES:
Drinking intentions | 4-weeks post-randomisation
  Change in next-month drinking intentions (5-point scale: 1, not at all; 5, to a very large extent)
Drinking intentions - standard drinks | 4-weeks post-randomisation
  Change in intended number of standard drinks consumed over the next month (composite of intention frequency/quantity response items)
Proportion of participants intending to reduce alcohol consumption | immediately post-randomisation
  Proportion of participants intending to reduce their next-month alcohol consumption (5-point scale: 1, not at all; 5, to a very large extent)
Proportion of participants intending to reduce alcohol consumption | 4-weeks post-randomisation
  Proportion of participants intending to reduce their next-month alcohol consumption (5-point scale: 1, not at all; 5, to a very large extent)
Knowledge of alcohol as a breast cancer risk factor | 4-weeks post-randomisation
  Proportion of participants accurately identifying alcohol as a clear risk factor for breast cancer
Alcohol literacy | 4-weeks post-randomisation
  Proportion of participants accurately identifying i) the increased breast cancer risk associated with drinking one average restaurant serve of wine a day; ii) the number of standard drinks in an average restaurant serve of red wine; iii) the maximum number of standard drinks per week recommended by current Australian Alcohol Guidelines (multiple-choice questions)
Alcohol consumption | 4-weeks post-randomisation
  Among women who have had an alcohol drink in the past month, change in alcohol consumption (composite of frequency/quantity response items)
Knowledge of other breast cancer risk factors | 4-weeks post-randomisation
  Proportion of participants accurately identifying inactivity and excess weight as risk factors for breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Jasmin Grigg, PhD, Principal Investigator — Turning Point, Eastern Health; Monash University
Locations (1):
- Maroondah BreastScreen, Ringwood East, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
There is not Ethics approval to seek patient permission to share data outside this study.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study Protocol containing summary Statistical Analysis Plan (2023-08-11): https://cdn.clinicaltrials.gov/large-docs/42/NCT06019442/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (Addendum) (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/42/NCT06019442/SAP_001.pdf